CLINICAL TRIAL: NCT00669825
Title: A Phase 1, Two Stage, Single-Blind, Single Dose, Placebo Controlled, Dose Escalation, Crossover Study of the Safety and Tolerability of ALV003 in Healthy Adult Volunteers and Subjects With Well-Controlled Celiac Disease Following a Gluten-Containing Meal
Brief Title: Study of ALV003 in Healthy Adult Volunteers and Subjects With Well-Controlled Celiac Disease Following a Gluten-Containing Meal
Acronym: FED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvine Pharmaceuticals Inc. (Industry)
Responsible Party: Vijaya Pratha, MD, Principal Investigator, Clinical Applications Laboratories Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ALV003-0812
Record Dates: First submitted 2008-04-21; First posted 2008-05-01 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Celiac Disease
Keywords: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — ALV003

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- B (Active Comparator): ALV003 (Active Study Drug)
  Interventions: Drug: ALV003

INTERVENTIONS:
Drug: ALV003 — Doses via intragastric tube at dosages of either 100 mg, 300 mg, 900 mg, or 1800 mg
  Arms: B
Drug: Placebo — Placebo to be administered via intragastric tube
  Arms: A

SUMMARY:
ALV003-0812 is a study of the safety and tolerability of a study drug (ALV003) in healthy adult volunteers and in patients with well-controlled celiac disease, following a meal that contains gluten.

DETAILED DESCRIPTION:
ALV003-0812 (the FED study) is designed to evaluate the safety and tolerability of a single dose of the study drug, ALV003, administered at one of four different dose levels, and following a test meal containing a small amount (1 gram) of gluten. ALV003 has been demonstrated to proteolyze (assist with the digestion of) various forms of gluten (gluten flour, wheat bread) in laboratory studies and in animals. Celiac disease has been estimated to affect 1% of the population of the United States, is related to gluten, and has a wide range of clinical manifestations including chronic gastrointestinal symptoms, malabsorption, and bone disease.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 45 years (inclusive)
* Healthy volunteers, in good health on the basis of medical history, physical examination, and laboratory values to include: hematology, chemistry, urinalysis, and liver function tests.
* Subjects with well-controlled celiac disease (CD), in good health with the exception of CD

  1. history of biopsy-proven CD in past 5 years
  2. on gluten free diet for at least 8 weeks prior to enrollment
  3. tTG or DGP titers within normal limits (≤ 15 IU)
  4. no flare in symptoms for the past 8 weeks
* Male or non-lactating, non-pregnant females who are postmenopausal, sterile or using at least two acceptable and highly effective birth control methods
* No systemic biologics may be taken for at least 6 months prior to Visit 2 and through 24 hours post-dose at Visit 3 Other than birth control, no prescribed medications, NSAIDs or aspirin may be taken for at least 7 days prior to Visit 2 and through 24 hours post-dose at Visit 3.
* No probiotics may be taken for at least 5 days prior to Visit 2 and through 24 hours post-dose at Visit 3.
* No over-the-counter medications and supplements may be taken for at least 3 days prior to Visit 2 and through 24 hours post-dose at Visit 3
* Body Mass Index of < 30 kg/m2
* Have understood and signed an Informed Consent Form
* Able and willing to comply with study requirements

Exclusion Criteria:

* Positive urine test for alcohol or illegal drugs at screening
* Positive breath test for Helicobacter pylori
* History (within the last 5 years) of inadequate acid secretion, either through a pentagastrin stimulated acid secretion test or fasting intragastric pH 2.5 or greater assessed by passage of a gastric pH probe in the fasting condition
* Aspirin or nonsteroidal anti-inflammatory drugs within 7 days prior to nasogastric or orogastric intubation at Visit 2
* The subject has received an experimental drug within 30 days
* History of substance abuse within the past 5 years
* Clinically significant abnormal lab values, as determined by the PI

  1. Liver Function Tests > 2.5 times Upper Limit of Normal (ULN)
  2. Serum Creatinine > 1.5 mg/dL
  3. Hemoglobin (Hb) < 10 g/dL
  4. Hematocrit outside of the normal range
  5. Platelet count < 150,000
  6. Serum Potassium, Prothrombin Time (PT), Partial Thromboplastin Time (PTT), or white blood cell count (WBC) outside of the normal range
* History of tobacco use within the last 6 months
* History of untreated or active peptic ulcer disease, esophagitis, motility disorders or any GI diseases in the past year
* Chronic use (more than once a week) of antacids, H2 receptor blockers or proton pump inhibitors
* Alcohol consumption of > 2 standard drinks equivalents per day
* Positive pregnancy test within 7 days prior to study drug administration
* Medical history (Healthy volunteers)

  1. gluten intolerance
  2. first degree relative diagnosed with celiac disease
  3. history of food allergies or digestive enzyme deficiencies
  4. history of any medically significant condition considered by PI to adversely affect participation
  5. chronic disease or condition
* Medical History (well-controlled CD subjects)

  1. history of any medically significant condition (other than CD) considered by PI to adversely affect participation
  2. chronic disease or condition other than CD
  3. history of severe reactions to low doses of gluten/accidental exposure to gluten
* History of a condition that is contraindicated for nasogastric or orogastric intubation
* Known allergy or hypersensitivity to any of the components of the test meal, placebo, study drug, E. coli-derived proteins or the 25% dextrose and water solution that will be used to flush the tube immediately following dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Throughout

CONTACTS AND LOCATIONS:
Overall Officials: Vijaya Pratha, MD, Principal Investigator — Clinical Applications Laboratories
Locations (2):
- United States (2):
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Clinical Applications Laboratories, San Diego, California